CLINICAL TRIAL: NCT02805452
Title: Impact of Solifenacin Succinate for Treatment of Acute Irritative Urinary Toxicity Occurring During Radiotherapy of Prostatic Cancer
Brief Title: Solifenacin Succinate for Treatment of Urinary Toxicity Occurring During Radiotherapy of Prostatic Cancer
Acronym: VesiCaP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Target of recruitment not reachable
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-RdC-PRO-Th; 2014-004296-22 (EudraCT Number)
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Succinate of Solifenacin (Experimental): 1 tablet of 5 mg of succinate of Solifenacin will be administered each day for 3 months.
  Interventions: Drug: Succinate of Solifenacin
- Placebo of Succinate of Solifenacin (Placebo Comparator): 1 tablet of placebo of succinate of solifenacin will be administered each day for 3 months.
  Interventions: Drug: Placebo of Succinate of Solifenacin

INTERVENTIONS:
Drug: Succinate of Solifenacin
  Arms: Succinate of Solifenacin
Drug: Placebo of Succinate of Solifenacin
  Arms: Placebo of Succinate of Solifenacin

SUMMARY:
The purpose of this study is to determine whether Succinate of Solifenacin reduces the OverActive Bladder syndrome occurring during prostate irradiation.

DETAILED DESCRIPTION:
A multicenter Phase III, randomized, double-blinded, parallel group placebo-controlled study.

2 groups:

* Control arm = pts. with placebo
* Experimental arm = pts. with Solifenacin succinate 5 mg - Vesicare® All patients with an OAB sub-score using the USP scale greater to 5 during prostate cancer radiotherapy will be included, receiving either a placebo or Solifenacin succinate (5mg) for duration of 3 months.

The randomization will be stratified on the radiotherapy dose (1 to 40 Gy or 40 to 70/80 Gy).

Screening:

For all patients, OAB items of the USP scale will be completed before each standard weekly assessment during prostate radiotherapy. Patients who reach an OAB sub-score greater to 5 will be addressed to an urologist in order to confirm absence of Qmax < 10ml/sec at initial assessment, or post-void residual urine > 100 milliliter (ml).

Inclusion & treatment:

A week at most after pre-screening, patients will be randomized to receive either Vesicare®-5mg or a placebo. In both study arms, the treatment should be continued for 3 months.

Follow-up:

The radiation oncologist will perform patients' follow-up for the study at the treatment initiation, 6 weeks and 3 months after start of the treatment (Vesicare or placebo).

The questionnaires for the evaluation of OAB syndrome, acute urinary toxicity and quality of life should be completed for each follow-up visit. The voiding diary will be completed during 3 days before (or if not, 3 days after) all the evaluation times.

An urologist will perform an uroflowmetry and a post-voiding echography (or a bladder scan) before initiation of the treatment, and after 6 weeks of treatment.

Statistics and sample size PATIENTS ENROLMENT 70 patients will be included (considering 66 patients completing the full study) within 3 recruitment centers

ELIGIBILITY:
Inclusion Criteria:

* Prostate adenocarcinoma (histological confirmation),
* Indication for prostate cancer radiotherapy (standard schema with a total dose from 70 to 80 Gray (GY)),
* Patient affiliation to the French Social Security System,
* Patient information and written informed consent,
* Patient complaining of urinary symptoms during radiotherapy,
* Occurrence of OverActive Bladder (OAB) subscore with the Urinary Symptom Profile (USP) scale greater or equal to 5.

Exclusion Criteria:

* Prostate irradiation contraindication
* History of bladder or prostate surgery,
* History of of pelvic radiotherapy,
* Individual deprived of liberty or placed Under the authority of a tutor,
* Age < 18 years,
* Flowmetry Qmax < 10ml/s and/or post-void residual urine > 100 ml (during urology preinclusion visit)
* Previous known OAB
* Patients treated with non-authorized drugs,
* Patients treated with anticholinergic or cholinesterase inhibitors within 12 months before irradiation,
* Patients treated with anticholinergic during and weeks following irradiation and before Succinate of Solifenacin treatment start,
* Patients treated with botulinum toxin within 9 months before screening,
* Patients treated with alpha-blockers, 5-alpha reductase inhibitor within 12 months preceding irradiation, during and weeks following irradiation and before Succinate of Solifenacin treatment start,
* Contraindication of Succinate of Solifenacin
* Hypersensitivity or allergy to Solifenacin succinate or to any other antimuscarinic agent,
* Specific precautions of use for patients having decompensated urinary tract obstruction at risk of urinary retention, vegetative neuropathy, long QT syndrome and an hypokaliemia, history of long QT or patients at risk of QT prolongation, obstructive gastrointestinal disorders.
* Patients treated with oral biphosphonates, drugs that cause QT prolongation or by substrates having affinity for CYP3A4 isoenzyme as verapamil and Diltiazem, or treated with CYP3A4 inductors as rifampicin, phenytoin, carbamazepine
* Galactose hereditary intolerance, lactase deficiency or a malabsorption syndrome of glucose and galactose.
* Patient enable to follow study medical care for family, social, geographical or psychological reasons.
* Participation to another clinical study on urinary toxicity and/or molecule that could modify this toxicity and its evolution.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Score of Urinary Symptom Profile (USP) questionnaire | At 6 weeks
  Score will be measured after study drug treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Crevoisier, MD, Principal Investigator — Centre Eugène Marquis
Locations (5):
- France (5):
  - Clinique Pasteur Lanroze, Brest
  - CH Bretagne Sud, Lorient
  - CH Lyon Sud, Lyon
  - Hôpital Saint Louis, Paris
  - Centre Eugene Marquis, Rennes

IPD SHARING:
Plan to Share IPD: No